CLINICAL TRIAL: NCT07144475
Title: Comparison of Probiotic Effects of Lactobacillus Casei Shirota With Lactobacillus Acidophilus on the Outcomes of Patients After Colorectal Cancer Surgery: A Study of Gastrointestinal Function, Sepsis Incidence, C-Reactive Protein, Interleukin 6 and Length of Stay
Brief Title: Comparison of Probiotic Effects on the Outcomes of Patients After Colorectal Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dharmais National Cancer Center Hospital (Other Government)
Responsible Party: Principal Investigator, Berial Dewin Marzaini, Principal Investigator, Dharmais National Cancer Center Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DP.04.03/11.7/020/2024
Record Dates: First submitted 2025-08-18; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: Probiotics; Lactobacillus casei Shirota; Lactobacillus acidophilus; Colorectal cancer; Surgical outcomes
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus casei Shirota Group (Active Comparator): Participants were given probiotic liquid beverage containing 6,5x10^9 CFU of Lactobacillus casei Shirota strain
  Interventions: Biological: Lactobacillus casei Shirota
- Lactobacillus acidophilus Group (Active Comparator): Participants were given Probiotic capsule containing 10^9 CFU of Lactobacillus acidophilus strain
  Interventions: Biological: Lactobacillus acidophilus

INTERVENTIONS:
Biological: Lactobacillus casei Shirota — Consumption of Lactobacillus casei Shirota three times daily for three days before surgery at 6 AM, 2 PM and 10 PM.
  Other Names: Yakult Light
  Arms: Lactobacillus casei Shirota Group
Biological: Lactobacillus acidophilus — Consumption of Lactobacillus acidophilus three times daily for three days before surgery at 6 AM, 2 PM and 10 PM.
  Other Names: Natrol Acidophilus Probiotic
  Arms: Lactobacillus acidophilus Group

SUMMARY:
This clinical trial aims to compare the effects of administering Lactobacillus casei Shirota probiotics with Lactobacillus acidophilus on the outcomes of patients after colorectal cancer surgery. Researchers will compare probiotic to see if Lactobacillus casei Shirota improves gastrointestinal function, sepsis incidence, C-reactive protein (CRP), interleukin 6 (IL-6), and length of stay better than Lactobacillus acidophilus. Participants will take probiotics three times daily for three days before surgery.

DETAILED DESCRIPTION:
The research design was a two-group unblinded, randomized clinical trial in 90 adult patients undergoing colorectal cancer surgery who are treated in the ICU, HCU and wards of Dharmais Cancer Hospital. Subjects who meet the criteria are divided into 2 (two) groups: the group given Lactobacillus casei Shirota and Lactobacillus acidophilus probiotics. Assessment of gastrointestinal function using the I-FEED score for early feeding was carried out on the second day after surgery. Sepsis diagnosis used the NEWS2 scoring assessed on the second, fourth, and sixth days of treatment. CRP levels were measured three times, namely during perioperative visit before surgery, four hours before surgery and three days after surgery. IL-6 levels were measured twice, namely perioperative visit before surgery and three days after surgery. Length of stay was calculated from after surgery until the patient was discharged.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed with colorectal cancer and would undergo resection surgery at Dharmais Cancer Hospital

Exclusion Criteria:

1. The patient or patient's family refused to be included in the study
2. Patients with chronic diseases such as HIV, uncontrolled diabetes mellitus (, uncontrolled cardiovascular disease and kidney failure
3. Patients with a history of regular probiotics, or steroids, or antibiotics consumption
4. Patients with anatomical disorders of the gastrointestinal system
5. Patients with immunocompromised conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Function | Second day of treatment in the ICU
  Assessed using I-FEED score which measures postoperative gastrointestinal function that contains five elements (intake, response to nausea treatment, emesis, examination, and duration, each scored with 0, 1, or 3 points) and classifies patients into normal, postoperative gastrointestinal intolerance (POGI), and postoperative gastrointestinal dysfunction (POGD)
Sepsis Incidence | second, fourth, and sixth days of treatment
  Assessed using NEWS2 to determine patient's degree of illness and prompts critical care intervention
C-reactive protein (CRP) | Baseline, four hours before surgery and three days after surgery
  CRP is a protein synthesized in the liver and will increase in response to inflammation. Baseline CRP data was collected on the same day the patient visited the oncology clinic before surgery and before probiotic consumption
Interleukin 6 (IL-6) | Baseline and three days after surgery
  IL-6 is a soluble mediator that has several functions in the immune response. IL-6 is produced in response to infection or tissue trauma. Baseline IL-6 data was collected on the same day the patient visited the oncology clinic before surgery and before probiotic consumption.
Length of stay | Up to 16 days (documented maximum length of stay)
  The number of days of patient care after undergoing colorectal cancer surgery until the patient can be treated as an outpatient

CONTACTS AND LOCATIONS:
Overall Officials: Berial D Marzaini, MD, Principal Investigator — Faculty of Medicine, University of Indonesia; Dita Aditianingsih, Professor, Study Chair — Faculty of Medicine, University of Indonesia; Arif HM Marsaban, MD, Study Chair — Faculty of Medicine, University of Indonesia; Gardian L Hakim, MD, Study Chair — Dharmais Cancer Hospital
Locations (1):
- Faculty of Medicine, University of Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arumugam S, Lau CS, Chamberlain RS. Probiotics and Synbiotics Decrease Postoperative Sepsis in Elective Gastrointestinal Surgical Patients: a Meta-Analysis. J Gastrointest Surg. 2016 Jun;20(6):1123-31. doi: 10.1007/s11605-016-3142-y. Epub 2016 Apr 12. PMID 27073082
- [Background] Khailova L, Frank DN, Dominguez JA, Wischmeyer PE. Probiotic administration reduces mortality and improves intestinal epithelial homeostasis in experimental sepsis. Anesthesiology. 2013 Jul;119(1):166-77. doi: 10.1097/ALN.0b013e318291c2fc. PMID 23571641
- [Background] Mulita F, Liolis E, Akinosoglou K, Tchabashvili L, Maroulis I, Kaplanis C, Vailas M, Panos G. Postoperative sepsis after colorectal surgery: a prospective single-center observational study and review of the literature. Prz Gastroenterol. 2022;17(1):47-51. doi: 10.5114/pg.2021.106083. Epub 2021 May 23. PMID 35371356
- [Background] Bai Y, Huang Y, Li Y, Zhang B, Xiao C, Hou X, Yu L. The Murine Reg3a Stimulated by Lactobacillus casei Promotes Intestinal Cell Proliferation and Inhibits the Multiplication of Porcine Diarrhea Causative Agent in vitro. Front Microbiol. 2021 Jun 18;12:675263. doi: 10.3389/fmicb.2021.675263. eCollection 2021. PMID 34220758
- [Background] Pak H, Maghsoudi LH, Soltanian A, Gholami F. Surgical complications in colorectal cancer patients. Ann Med Surg (Lond). 2020 May 11;55:13-18. doi: 10.1016/j.amsu.2020.04.024. eCollection 2020 Jul. PMID 32435475
- [Background] Shida K, Kiyoshima-Shibata J, Nagaoka M, Watanabe K, Nanno M. Induction of interleukin-12 by Lactobacillus strains having a rigid cell wall resistant to intracellular digestion. J Dairy Sci. 2006 Sep;89(9):3306-17. doi: 10.3168/jds.S0022-0302(06)72367-0. PMID 16899663
- [Background] Alsharqawi N, Alhashemi M, Kaneva P, Baldini G, Fiore JF Jr, Feldman LS, Lee L. Validity of the I-FEED score for postoperative gastrointestinal function in patients undergoing colorectal surgery. Surg Endosc. 2020 May;34(5):2219-2226. doi: 10.1007/s00464-019-07011-6. Epub 2019 Jul 30. PMID 31363895
- [Background] Tan CK, Said S, Rajandram R, Wang Z, Roslani AC, Chin KF. Pre-surgical Administration of Microbial Cell Preparation in Colorectal Cancer Patients: A Randomized Controlled Trial. World J Surg. 2016 Aug;40(8):1985-92. doi: 10.1007/s00268-016-3499-9. PMID 27098538
- [Background] Pitsillides L, Pellino G, Tekkis P, Kontovounisios C. The Effect of Perioperative Administration of Probiotics on Colorectal Cancer Surgery Outcomes. Nutrients. 2021 Apr 25;13(5):1451. doi: 10.3390/nu13051451. PMID 33922897
- [Background] Qin D, Ma Y, Wang Y, Hou X, Yu L. Contribution of Lactobacilli on Intestinal Mucosal Barrier and Diseases: Perspectives and Challenges of Lactobacillus casei. Life (Basel). 2022 Nov 16;12(11):1910. doi: 10.3390/life12111910. PMID 36431045
- [Background] Dempsey E, Corr SC. Lactobacillus spp. for Gastrointestinal Health: Current and Future Perspectives. Front Immunol. 2022 Apr 6;13:840245. doi: 10.3389/fimmu.2022.840245. eCollection 2022. PMID 35464397